CLINICAL TRIAL: NCT03479346
Title: Exploring the Efficacy and Safety of Herbal Medicine on Korean Obese Women With or Without Metabolic Syndrome Risk Factors - A Study Protocol for a Double-blind, Randomised, Multi-center, Placebo-controlled Clinical Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gachon University Gil Oriental Medical Hospital (Other)
Collaborators: DongGuk University (Other); Wonkwang University Guangju Medical Center (Unknown); Dongsin University Oriental Hospital (Unknown); Kyunghee University Medical Center (Other)
Responsible Party: Principal Investigator, Yun-Kyung Song, Principal investigator, Gachon University Gil Oriental Medical Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ISEE_2017_GGT
Record Dates: First submitted 2018-03-21; First posted 2018-03-27 (Actual); Last update posted 2021-04-12 (Actual); Status verified 2021-04

CONDITIONS: Obesity; Metabolic Syndrome
Keywords: Obesity; Metabolic syndrome; Traditional Korean Medicine; Galgeun-tang
MeSH Terms: conditions — Obesity; Metabolic Syndrome | interventions — galgeun-tang

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GGT group (Experimental): Usage: 3g, three times a day, each taken before or between meals for 12 weeks Manufacturing company: HANPOONG PHARM & FOODS Co. Ltd.
  Interventions: Drug: GGT
- Placebo group (Placebo Comparator): Usage: 3g, three times a day, each taken before or between meals for 12 weeks Manufacturing company: HANPOONG PHARM & FOODS Co. Ltd.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: GGT — Usage: 3g, three times a day, each taken before or between meals for 12 weeks Manufacturing company: HANPOONG PHARM & FOODS Co. Ltd.
  Other Names: Galgeun-tang
  Arms: GGT group
Drug: Placebo — Usage: 3g, three times a day, each taken before or between meals for 12 weeks Manufacturing company: HANPOONG PHARM & FOODS Co. Ltd.
  Arms: Placebo group

SUMMARY:
The Purpose of this trial is to investigate the efficacy and safety of GGT on Korean obese Women with or without metabolic syndrome Risk factors

ELIGIBILITY:
Inclusion Criteria:

* Female aged 19 to 65 years

  * Subject must included at least one or more of the following symptoms below;

    * BMI of 30 kg/㎡ or more;
    * BMI between 27 and 29.9kg/㎡ with non-insulin-dependent diabetes mellitus, taking medication or fasting blood glucose > 126mg/dL at the screening visit
    * BMI between 27 and 29.9kg/㎡ with hyperlipidemia, taking medication or total cholesterol ≥ 200mg/dL or Triglyceride ≥ 150mg/dL at screening visit
* Agreed to low-calorie diet during the trial
* Written informed consent of the trial

Exclusion Criteria:

* Subjects who had experience with allergic reaction on investigational drug(any ingredients of IP)

  * Subjects who has diabetes as comorbidity, had experienced the elevation of blood glucose by ephedrine
  * Subjects who had experienced rash, rubefaction, or itchiness by GGT administration
  * Subjects who usually feel fatigue due to hyperhidrosis
  * Subjects who experienced other allergic reactions
* Subjects who had 10 percent reduction in body weight over 6 months
* Subjects who decided to quit smoking over the last 3 months or have irregular smoking habits
* Subjects who have endocrine diseases associated with weight gain, such as hypothyroidism, Cushing's syndrome, etc.
* Subjects who have heart disease (heart failure, angina pectoris, myocardial infarction)
* Subjects who have uncontrolled hypertension despite the use of antihypertensive drugs (SBP > 145 mmHg or DBP > 95 mmHg)
* Subjects who have uncontrolled diabetes despite the use of drugs (FBS>7.8 mmol/L (140 mg/dL))
* Subjects who have severe renal disability (SCr > 2.0 mg/dL)
* Subjects who have severe liver disability (2.5 fold of normal high range value on Alanine Aminotransferase [ALT], Aspartate Aminotransferase [AST], alkaline phosphatase [ALP])
* Subjects who have poor digestion(anorexia, stomach discomfort, nausea, vomiting etc) or have the history of eating disorder such as anorexia nervosa or bulimia nervosa, etc.(KEAT-26 < 20)
* Use of medication that can affect on weight within last 3 months (appetite suppressant, laxative, oral steroid, thyroid hormone, amphetamine, cyproheptadine, phenothiazine or medications can affect on absorption, metabolism, excretion)
* Use of CNS stimulant medication for weight loss
* Subjects who had a use of drugs that can increase blood pressure or heart rate within a week, such as, Decongestants, cough, cold, allergy treatments that include the ingredients of phenylpropanolamine, ephedrine, pseudoephedrine
* Forbidden treatment (Insulin, hypoglycemic agent, antidepressant, antiserotonin agent, barbiturate, antipsychotic, medication concerns of abuse)
* Subjects who have diseases that may occur hypokalemia (hypomagnesemia, Bartter syndrome, Gitelman syndrome, diseases that can cause high aldosteronism etc.) or have cardiac dysrhythmia
* Difficult to measure anthropometric dimensions because of anatomical change such as resection
* History of weight loss surgery, such as bariatric surgery, etc.
* Edema or dysuria
* Malignant tumour or lung disease
* Cholelithiasis
* History of narrow angle glaucoma
* Subjects who have nervous or psychological medical history or presently suffer from the following diseases: depression, manic disorder, bipolar disorder, schizophrenia, epilepsy, alcoholism, anorexia, hyperphagia, etc.
* Subjects who have history of stroke or temporary ischemic cardioplegia
* Subjects who are judged to be inappropriate for the clinical study by the researchers
* Women who were pregnant, lactating or have the chances of pregnancy who do not agree to proper contraception (birth-control pill, hormone implant, IUD, spermicide, condom, abstinence, etc.)
* Use of other investigational product within last 1 month

Ages: 19 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2018-04-28 (Actual); Primary Completion 2020-10-01 (Actual); Study Completion 2020-12-01 (Actual)

PRIMARY OUTCOMES:
Changes from baseline in body weight | baseline, 12 weeks
  Estimated mean changes from baseline in body weight after 12 weeks of treatment.

SECONDARY OUTCOMES:
Changes from baseline in body fat percentage | baseline, 4,8,12 weeks
  Estimated mean changes from baseline in body fat percentage at different time points during treatment period
Changes from baseline in fat mass | baseline, 4,8,12 weeks
  Estimated mean changes from baseline in fat mass at different time points during treatment period
Changes from baseline in Waist circumference | baseline, 4,8,12 weeks
  Estimated mean changes from baseline in Waist circumference at different time points during treatment period
Changes from baseline in Waist/hip ratio | baseline, 4,8,12 weeks
  Estimated mean changes from baseline in Waist/hip ratio at different time points during treatment period
Changes from baseline in Body mass index | baseline, 4,8,12 weeks
  Estimated mean changes from baseline in Body mass index at different time points during treatment period
Changes from baseline in Lipid profile | Screening visit, 12 weeks
  Estimated mean changes from first visit in Lipid profile after 12 weeks of treatment.
Changes from baseline in C-reactive protein (CRP) | baseline, 12 weeks
  Estimated mean changes from baseline in C-reactive protein (CRP) after 12 weeks of treatment.
Changes from baseline in blood glucose | Screening visit, 12 weeks
  Estimated mean changes from first visit in blood glucose after 12 weeks of treatment.
European Quality of life 5 Dimension(EQ5D) | baseline, 12 weeks
  EQ-5D is a tool developed for health-related quality of life (HRQoL) assessment, and is widely used in the health care sector. Scores range from -1, 'health worse than death' to 1, 'perfect health'. EQ-5D-5L has 5 dimensions covering current health status and functionality: mobility (M), self care (SC), usual activities (UA), pain/discomfort (PD), and anxiety/depression (AD), to be rated out of 5 grades (1, no problem; 2, slight problem; 3, some/moderate problem; 4, severe problem; 5, extreme problem).
Changes from baseline in serum leptin | baseline, 12 weeks
  Estimated mean changes from first visit in serum leptin after 12 weeks of treatment.
Korean version of Western Ontario and McMasters Universities Oateoarthritis Index | baseline, 12, 16 weeks
  Determination of patient's knee function and pain
cost per QALY(Quality Adjusted Life Years) gained | 6 months or 1 year
  The cost per QALY gained is calculated according to normal health-economic evaluation models.
Economic evaluation (medical costs) | baseline, 4,8,12,16,20,24 weeks
  Economic evaluation of medical costs will be performed to assess cost-effectiveness of the 2 groups.
Economic evaluation (time-related costs) | baseline, 4,8,12,16,20,24 weeks
  Economic evaluation of time-related costs will be performed to assess cost-effectiveness of the 2 groups.
Economic evaluation (lost productivity costs) | baseline, 4,8,12,16,20,24 weeks
  Economic evaluation of lost productivity costs will be performed to assess cost-effectiveness of the 2 groups.

OTHER OUTCOMES:
Changes from baseline in Kellgren-Lawrence grade | baseline, 12 weeks
  Determination of patient's knee condition

CONTACTS AND LOCATIONS:
Overall Officials: Yun-Kyung Song, PhD, Principal Investigator — Gachon University Gil Oriental Medical Hospital
Locations (1):
- Gachon University Gil Oriental Medical Hospital, Incheon, South Korea

IPD SHARING:
Plan to Share IPD: No